CLINICAL TRIAL: NCT07404007
Title: Detection of Proximal Caries in Bitewing Radiography Using Artificial Intelligence - A Diagnostic Clinical Study
Brief Title: Detection of Proximal Caries in Bitewing Radiography Using Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, Associate Professor, Conservative dentistry department, Cairo University
Other Study IDs: CONS_ Rad 1180
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Proximal Caries; Tooth Caries
Keywords: Artificial intelligence; Proximal caries; A Diagnostic accuracy Study
MeSH Terms: conditions — Dental Caries | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Group 1 Artificial Intelligence Deep learning that is applied in Diagnosis of the proximal Caries
  Interventions: Diagnostic Test: Artificial Intelligence (AI): Deep learning that is applied in Diagnosis of the proximal Caries
- Group 2 : Digital Bitewing manually annotated by human experts
  Interventions: Diagnostic Test: Manual annotation of Digital Bitewing Radiograph by human experts

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence (AI): Deep learning that is applied in Diagnosis of the proximal Caries — Artificial intelligence was used as a deep-learning diagnostic tool to detect proximal caries on digital bitewing radiographs. The system analyzed images and generated probability scores and visual markers for suspected lesions. Its performance was compared with expert examiner diagnoses as the reference standard. AI results were used for evaluation only and did not influence patient treatment decisions.
  Groups: Group 1 Artificial Intelligence Deep learning that is applied in Diagnosis of the proximal Caries
Diagnostic Test: Manual annotation of Digital Bitewing Radiograph by human experts — Digital bitewing radiographs were manually annotated by calibrated human experts to identify the presence and location of proximal caries. Annotations were performed using standardized diagnostic criteria and dedicated imaging software to mark suspected lesions. These expert markings served as the reference standard for comparison with the artificial intelligence outputs. Inter-examiner agreement was assessed, and disagreements were resolved by consensus.
  Groups: Group 2 : Digital Bitewing manually annotated by human experts

SUMMARY:
Using a sequence of bitewing radiographs, Artificial intelligence assists in identifying interproximal caries. For the identification of dental caries in bitewing, periapical, and panoramic radiographs, a trained deep learning network will be created This study aimed to investigate the reliability of a novel Artificial Intelligence model based on deep learning in the detection of Proximal Caries using Digital Bitewing Radiographs. (BW).

ELIGIBILITY:
Inclusion Criteria:

* Patients having all Permanent premolars and molars (maximum one tooth missing on each side)

Exclusion Criteria:

* 1-Dental Anomalies →Amelogenesis Imperfecta, Dentinogenesis Imperfecta, taurodontism 2- Severe crowding which prevent visualization of teeth Contacts 3-Orthodontic wires bonded to Enamel of the tooth

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Faculty dental out patient clinic who required bitewing radiographic examination for routine diagnosis or treatment planning.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Reliability of the artificial intelligence model in detecting proximal caries on digital bitewing radiographs | cross-sectional assessment at baseline, with no follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No